CLINICAL TRIAL: NCT00004071
Title: A Randomized, Open-Label Phase II/III Study of SU101 Plus Mitoxantrone/Prednisone Compared to Mitoxantrone/Prednisone Alone in Patients With Hormone-Refractory Prostate Cancer
Brief Title: Mitoxantrone and Prednisone With or Without Leflunomide in Treating Patients With Stage IV Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SUGEN-SU101.035; CDR0000067275; SUGEN-990711
Record Dates: First submitted 1999-12-10; First posted 2004-06-04 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leflunomide; Mitoxantrone; Prednisone

INTERVENTIONS:
Drug: leflunomide
Drug: mitoxantrone hydrochloride
Drug: prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if mitoxantrone and prednisone are more effective with or without leflunomide for treating prostate cancer.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of mitoxantrone and prednisone with or without leflunomide in treating patients who have stage IV prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the percentage one year survival rate in hormone refractory prostate cancer patients treated with leflunomide (SU101), mitoxantrone, and prednisone versus mitoxantrone and prednisone alone. II. Compare the palliative pain response, time to treatment failure, time to progression, median survival, investigator global response assessment, objective response, time to palliative pain response, duration of palliation, and effect on PSA between these two regimens. III. Assess the safety and tolerability of mitoxantrone in combination with SU101 in these patients. IV. Assess the health related quality of life of these patients on these regimens.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified by performance status (70-80% vs 90-100%), baseline present pain intensity score (2.0 vs greater than 2.0), and hemoglobin level (less than 12.0 g/dL vs at least 12.0 g/dL). Patients enter one of two treatment arms: Arm I: Patients are premedicated with an IV 5-HT3 reuptake inhibitor (i.e., odansetron) then receive mitoxantrone IV on day 1. Twice daily oral prednisone therapy begins on day 1 and continues throughout study treatment. Treatment repeats every 21 days for 4 courses. Arm II: Patients are premedicated with an IV 5-HT3 reuptake inhibitor as in arm I. Patients receive mitoxantrone and prednisone therapy as in arm I. Additionally, beginning on day 1 patients receive leflunomide (SU101) IV over 4-5 hours weekly for 12 weeks. The SU101 infusions shall precede mitoxantrone infusions. Patients receive a maximum of one year therapy with SU101; mitoxantrone therapy may be administered up to a maximum dose of 140/m2. Quality of life is assessed at baseline, day 8, day 21, and then every 3 weeks thereafter until study completion. Patients are followed at least every 2 months.

PROJECTED ACCRUAL: Up to 370 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hormone refractory stage IV prostate cancer Hormone refractory disease is defined as: Progressive measurable disease OR Progressive disease by bone scan OR Increase in PSA by 50% over nadir level confirmed twice and measured at least two weeks apart Prior treatment with primary androgen ablative therapy with castrate levels of testosterone Minimum score of 2 on the McGill 6 point pain scale secondary to metastatic bony pain with an analgesic score of at least 4 No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Greater than 16 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.0 g/dL (without blood transfusion(s) within 2 weeks prior to study) Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) AST no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No cardiac failure No myocardial infarction within the past 6 months No uncontrolled hypertension LVEF greater than 50% Other: Fertile patients must use effective barrier contraception during and for 3 months after study No known hypersensitivity to polysorbate or polyethylene glycol No other malignancies within past 5 years, except basal cell skin cancer No other acute or chronic medical, psychiatric, or lab abnormality that would prevent compliance No uncontrolled peptic ulcer No active infection No contraindication to mitoxantrone therapy No contraindication to prednisone therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic response modifiers At least 4 weeks since prior immunotherapy No concurrent immunotherapy Chemotherapy: No prior SU101 or mitoxantrone No prior cytotoxic chemotherapy for prostate cancer No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 4 weeks since prior antiandrogen therapy and recovered Concurrent primary androgen ablation therapy (orchidectomy, luteinizing hormone releasing hormone (LHRH) agonist (if stable dose), estrogen, or cyproterone acetate) allowed No concurrent antiandrogen therapy (except LHRH) No concurrent cholestyramine Radiotherapy: At least 4 weeks since prior radiotherapy (8 weeks since strontium 89 and samarium 153) Prior palliative radiotherapy to metastatic sites allowed No prior radiotherapy to greater than 50% of bone marrow No concurrent radiotherapy except for palliation of bone pain Surgery: At least 2 weeks since prior major surgery No concurrent surgery for prostate cancer Other: At least 4 weeks since prior investigational therapy At least 4 weeks since prior antiangiogenesis therapy At least 6 weeks since prior bicalutamide No other concurrent investigational therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack H. Mabry, MD, Study Chair — SUGEN
Locations (3):
- United States (3):
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - St. Vincents Comprehensive Cancer Center, New York, New York